CLINICAL TRIAL: NCT05957575
Title: Comparison of the Muscle Oxygenation During Submaximal and Maximal Exercise Tests in Patients With Post COVID-19 Syndrome
Brief Title: Investigation of the Muscle Oxygenation in Patients With Post COVID-19 Syndrome
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Other Study IDs: Gazi University 5
Record Dates: First submitted 2023-07-21; First posted 2023-07-24 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: COVID-19; oxygen consumption
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
More than 60% of patients infected with COVID-19 have long-term symptoms. These symptoms are associated with common ground-glass opacities on computed tomography scans and chest radiographs. The pathophysiology of long-term persistent symptoms is largely unknown, but hypoxia and hypoxic tissue damage, decreased pulmonary diffusion capacity, ventilation-perfusion mismatch, and lung fibrosis caused by COVID-19-associated pneumonia are thought to cause long-term symptoms. Desaturation may occur during exercise due to hypoxia, pneumonia and lung involvement in patients with post-COVID syndrome. Oxygenation of peripheral muscles may decrease due to hypoxemia, but there is not enough study on this subject yet.

DETAILED DESCRIPTION:
Post-COVID syndrome is defined as unexplained signs or symptoms that develop during or after infection with COVID-19 and persist for 12 weeks. Long-term symptoms include fatigue, dyspnea, impaired exercise and lung function.It is important to understand physiological mechanisms underlying persistent dyspnea, fatigue, and impaired exercise capacity after COVID-19 infection to develop appropriate rehabilitation interventions while improving these symptoms. The pathophysiology of long-term persistent symptoms is largely unknown, however hypoxia and hypoxic tissue damage caused by COVID-19-associated pneumonia, decreased pulmonary diffusion capacity, ventilation-perfusion mismatch and lung fibrosis have been hypothesized. The effect of hypoxemia associated with COVID-19 on oxygenation of peripheral muscles and muscle oxygenation at submaximal and maximal exercise intensity has not been investigated, yet.

The aim of our study is to evaluate and compare quadriceps femoris muscle oxygenation in submaximal and maximal exercise tests in patients with post-COVID syndrome.

Patients referred from Gazi University, Faculty of Medicine, Department of Chest Diseases for pulmonary rehabilitation to Cardiopulmonary Rehabilitation Unit located in the Faculty of Health Sciences were recruited, Department of Physiotherapy and Rehabilitation, between March 2022 and May 2023. Muscle oxygenation during six-minute walk test and cardiopulmonary exercise test on two different days was measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75
* Diagnosed with pulmonary involvement COVID-19
* Volunteer to participate in the study

Exclusion Criteria:

* Body mass index >35 kg/m2
* Acute pulmonary exacerbation, acute upper or lower respiratory tract infection
* Aortic stenosis, complex arrhythmia, aortic aneurysm
* Serious neurological, neuromuscular, orthopedic, other systemic diseases or other diseases affecting physical functions
* Cognitive impairment that causes difficulty in understanding and following exercise test instructions
* Participated in a planned exercise program in the last three months
* Uncontrolled hypertension and/or diabetes mellitus, heart failure and cardiovascular disease
* Contraindication for exercise testing and/or exercise training according to the American College of Sports Medicine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty eight patients with pulmonary involvement post-COVID syndrome were recruited for the study. Pulmonary involvement of the patients was determined by a pulmonologist according to the results of computed tomography.Patients referred from Gazi University, Faculty of Medicine, Department of Chest Diseases for pulmonary rehabilitation to Cardiopulmonary Rehabilitation Unit located in the Faculty of Health Sciences were recruited, Department of Physiotherapy and Rehabilitation.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Measurement of muscle oxygenation (SmO2) | through study completion, an average of 18 months
  The saturation of oxygen in muscles (SmO2) was evaluated using a non-invasive method Moxy® device (Moxy®, Fortiori Design LLC, Minnesota, USA).

SECONDARY OUTCOMES:
Maximal exercise capacity | through study completion, an average of 18 months
  Cardiopulmonary Exercise Test
Submaximal exercise capacity | through study completion, an average of 18 months
  Six minute walk test
Peripheral Muscle Strength | through study completion, an average of 18 months
  Hand held dynamometer
Functional Status | through study completion, an average of 18 months
  Post-COVID-19 Functional Status scale (PCFS)

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, Pt. MSc., Principal Investigator — Gazi University; Ece BAYTOK, Pt. MSc., Principal Investigator — Gazi University; Nilgün YILMAZ DEMİRCİ, Assoc. Prof., Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No